CLINICAL TRIAL: NCT07328399
Title: Impact of COVID-19 Pandemic Waves on Colorectal Cancer Stage Migration and Diagnostic Delays
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: IG/2037-1/2023
Record Dates: First submitted 2025-12-14; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: COVID-19; colorectal cancer; pandemic waves; follow-up
MeSH Terms: conditions — Colorectal Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Patients with colorectal cancer undergoing MRI examination during and after the COVID-19 pandemic.

SUMMARY:
Background/Objectives: The incidence of colorectal cancer in Hungary exceeds the EU (European Union) average, and the cancer mortality rate is also among the highest in the country. The COVID-19 pandemic has impacted various areas of healthcare, including cancer diagnosis and treatment. Due to the measures taken to combat the COVID-19 pandemic, not only newly suspected cancer patients but also those already diagnosed and undergoing treatment faced numerous difficulties. Methods: The study included 198 patients with colorectal cancer, of whom 43 participants were newly diagnosed cases. Due to low case numbers in certain COVID-19 waves, adjacent waves were merged for statistical analysis. The number of newly diagnosed colorectal cancer cases across COVID-19 waves was compared using one-way ANOVA, stage distribution differences and the proportion of missed treatments were assessed with Fisher's exact test. In follow-up patients, changes were analyzed using the Wilcoxon signed-rank test. Differences in tumor size categories were examined using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or confirmed colorectal cancer
* Patients examined by MRI at Szent Margit Hospital
* MRI referral issued between September 2020 and December 2023

Exclusion Criteria:

* MRI referrals not issued by Szent Margit Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with colorectal cancer undergoing MRI examination during and after the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Tumor stage distribution across COVID-19 pandemic waves | September 2020 - December 2023
  Comparison of colorectal cancer tumor stage (AJCC 8th edition) across different COVID-19 pandemic waves and the post-COVID period based on MRI findings.
Number of newly diagnosed colorectal cancer cases | September 2020 - December 2023
  Monthly number of newly diagnosed colorectal cancer cases across COVID-19 waves and the post-COVID period.
TNM classification | September 2020 - December 2023
  TNM classification of colorectal cancer according to the AJCC 8th edition during different COVID-19 pandemic waves in newly diagnosed and follow-up patients.

SECONDARY OUTCOMES:
Tumor progression or regression in follow-up patients | September 2020 - December 2023
  Change in tumor stage between previous imaging and most recent MRI examination.
Missed oncologic treatments | September 2020 - December 2023
  Occurrence of missed or delayed oncologic treatments documented during the COVID-19 pandemic period.
Presence and distribution of metastases | September 2020 - December 2023
  Presence, number, and organ distribution of metastatic disease based on imaging findings.

CONTACTS AND LOCATIONS:
Overall Officials: József Tollár, Dr., Principal Investigator — University of Pécs, Faculty of Health Sciences, Hungary; Adrienn Biró, Dr., Principal Investigator — Somogy County Móricz Kaposi Teaching Hospital, 7400 Kaposvár, Hungary
Locations (1):
- Szent Margit Hospital, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No